CLINICAL TRIAL: NCT00832507
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Multicenter, Dose-ranging Study of Cicletanine in Subjects With Pulmonary Arterial Hypertension
Brief Title: Study of Cicletanine for Pulmonary Arterial Hypertension (PAH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-235-0101
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; pulmonary hypertension; cicletanine; cicletanine HCL; cardiovascular; endothelin receptor antagonist; ERA; monotherapy; combination therapy; phosphodiesterase type-5 inhibitor; PDE5i; parenteral prostanoid; PH; pulmonary
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — cicletanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cicletanine 150 mg QD (Experimental): Cicletanine 150 mg administered once daily (QD)
  Interventions: Drug: Cicletanine
- Cicletanine 150 mg BID (Experimental): Cicletanine 150 mg administered twice daily (BID)
  Interventions: Drug: Cicletanine
- Cicletanine 300 mg QD (Experimental): Cicletanine 300 mg administered once daily (QD)
  Interventions: Drug: Cicletanine
- Placebo (Placebo Comparator): Placebo to match cicletanine administered once daily
  Interventions: Drug: Cicletanine; Drug: Cicletanine Placebo

INTERVENTIONS:
Drug: Cicletanine — Cicletanine capsules 150 mg or 300 mg administered orally once or twice daily
Drug: Cicletanine Placebo — Placebo to match cicletanine administered orally once daily, followed by active cicletanine in the blinded extension period
  Arms: Placebo

SUMMARY:
This Phase 2, randomized, double-blind, placebo-controlled, multicenter, dose-ranging study will compare the efficacy, safety, and tolerability of cicletanine hydrochloride (HCl) to placebo in subjects with PAH. Study drug will be administered alone, or on the background of stable PAH therapy. The study will consist of 3 periods: a screening period, a 12-week placebo-controlled treatment period, and a long-term, blinded extension period.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the change in exercise capacity following treatment with cicletanine HCl or placebo in subjects with PAH.

The secondary objectives of this study are:

1. To compare the change in other clinical measures of PAH following treatment with cicletanine HCl or placebo in subjects with PAH
2. To compare the safety and tolerability of cicletanine HCl to placebo in subjects with PAH Additionally, the long-term safety, tolerability, and efficacy of cicletanine HCl treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria

* Between 16 and 70 years of age
* Weigh greater than or equal to 40 kg
* Have a current diagnosis of IPAH, FPAH, or PAH that is primarily due to: connective tissue disease, congenital heart defects, drug and toxin use, and HIV infection
* Meet all of the following hemodynamic criteria by means of a RHC completed prior to or during Screening: mPAP of greater than or equal to 25 mmHg, PVR greater than 240 dyne.sec/cm5, PCWP or LVEDP of less than or equal to1 5 mmHg
* Walk a distance of at least 100 m but no more than 450 m during the screening 6MWT
* Have WHO functional class II, III, or IV symptoms
* Meet all of the following pulmonary function tests completed no more than 12 weeks before the Screening visit: TLC greater than or equal to 60% of predicted normal & FEV1 greater than or equal to 65% of predicted normal, FEV1:FVC ratio greater than 0.60
* Have laboratory results within 90% of the lower limit of normal to 1.5 times the upper limit of normal
* Receiving treatment with an approved ERA, PDE5i, and/or parenteral prostanoid must be receiving this therapy for greater than or equal to 12 weeks prior to the Screening Visit and must be at a stable dose for greater than or equal to 4 consecutive weeks prior to the Screening Visit.
* Eligible therapies allowed at Screening include:a. Monotherapy with an ERA, PDE5i, or parenteral prostanoid that is approved for the treatment of PAH b. Combination therapy with two eligible PAH treatments (any combination of ERA, PDE5i, or parenteral prostanoid
* Subject receiving diuretic treatment must be on stable therapy
* If receiving digitalis, CCBs, angiotensin receptor blockers (ARBs), angiotensin converting enzyme (ACE) inhibitors, or beta-blocking agents subject must be on stable therapy
* If receiving HMG-CoA reductase inhibitors, subject must be on stable therapy
* If diagnosis of HIV subject must have stable disease status
* Female subjects of childbearing potential must have a negative serum pregnancy test
* Female subjects of childbearing potential must agree to use 2 reliable methods of contraception
* Must agree not to participate in a clinical study involving another investigational drug or device
* Must be competent to understand and sign the IRB approved ICF
* Has not enrolled in an exercise training program for pulmonary rehabilitation and must agree not to enroll in an exercise training program for pulmonary rehabilitation
* If subject has been enrolled in an exercise training program for pulmonary rehabilitation for greater than 12 weeks prior to the Screening Visit and must agree to maintain their current level of rehabilitation for the first 12 weeks of the study
* Must be on background PAH therapy at Screening unless the subject does not have access to or can not tolerate currently approved PAH medical therapies

Exclusion Criteria

* Subject with a current PH diagnosis other than IPAH, FPAH, or PAH that is primarily due to: Connective tissue disease, Congenital heart defects, Drug and toxin use, or HIV infection
* Subject with LVEF less than or equal to 40% or clinically significant ischemic, valvular, or constrictive heart disease
* Subject with WHO functional class I symptoms
* Subject has chronically received an ineligible PAH treatment regimen within the 4 weeks prior to the Screening Visit, specifically: a. inhaled iloprost or inhaled treprostinil, b. combination treatment with three PAH therapies, c.any investigational therapy for the treatment of PAH d.Chronic use is considered greater than 7 consecutive days of treatment
* Subject receiving iv inotropes within 2 weeks prior to the Screening Visit
* Subject with SBP greater than or equal to 150 mmHg or less than 90mmHg
* Subject with moderate to severe liver disease
* Subject with moderate or severe renal impairment
* Subject receiving lithium within the 2 weeks prior to the Screening Visit
* Subject requiring intermittent or chronic treatment with nitrates
* Subject receiving non-anti-arrhythmic drugs
* Subject has a diagnosis of long QT syndrome
* Subject with evidence of chronic thromboembolic disease
* Subject with obstructive lung disease
* Subject with severe arthritis, musculoskeletal problems, or morbid obesity that would affect the subject's ability to perform or complete the 6MWT
* Has a history of malignancies within the past 5 years
* Subject with disease that may adversely affect the safety of the subject and/or efficacy of the study drug or severely limit the lifespan of the subject
* Female subject who is pregnant or breastfeeding
* Has demonstrated noncompliance with previous medical regimens
* Has a recent history of abusing alcohol or illicit drugs
* Has participated in a clinical study involving another investigational drug or device within 4 weeks before the Screening Visit
* Has a known hypersensitivity to the study drug, the metabolites, or formulation excipients
* Receiving an oral arginine supplement within 2 weeks prior to the Screening Visit

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in six-minute walk distance (6MWD) evaluated after 12 weeks of treatment | Baseline to Week 12

SECONDARY OUTCOMES:
Change from baseline in BDI, WHO Functional Class, BNP, cardiac hemodynamics and SF-36 physical functioning scale following 12 weeks of treatment. In addition, time to clinical worsening (TTCW) will be evaluated. | Baseline to Week 60

CONTACTS AND LOCATIONS:
Overall Officials: Gennyne Walker, PhD, Study Chair — Senior Clinical Research Scientist, Gilead Sciences
Locations (56):
- United States (39):
  - University of South Alabama, Mobile, Alabama
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - VA Greater LA Healthcare System, Los Angeles, California
  - University of California San Diego Medical Center, San Diego, California
  - Harish H. K. Murthy, MD, San Jose, California
  - UCLA Medical Center, Torrance, California
  - University of Colorado Denver, Aurora, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Cleveland Clinic, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - University of Chicago Hospital, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Louisiana State University, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Beth Israel Medical Center, New York, New York
  - Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - Case Medical Center, Cleveland, Ohio
  - Davis Heart and Lung Research Institute, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University Of Virginia, Charlottesville, Virginia
- Australia (2):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Royal Perth Hospital, Perth, Western Australia
- Austria (2):
  - University Klinik Graz, Graz
  - University Klinik Wien, Vienna
- ULB Hôpital Erasme, Brussels, Belgium
- Canada (3):
  - Peter Lougheed Centre, Calgary, Alberta
  - London Health Sciences Centre, London, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Germany (2):
  - Ludwig-Maximilians-Universitaet, Munich, Bavaria
  - Universitaetsklinikum Giessen und Marburg, Giessen, Hesse
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
- Mexico (2):
  - Unidad de Investigación Clínica en Medicina S.C., Monterrey, Nuevo León
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City
- Spain (2):
  - H Clinic i Provincial, Barcelona
  - HU 12 de Octubre, Madrid
- Royal Free Hospital, London, Gt Lon, United Kingdom